CLINICAL TRIAL: NCT06298357
Title: Virtual Reality Gaming for Exercise and Mindfulness Among Pediatric Cancer Rehabilitation Patients: Pilot Randomized Controlled Trial
Brief Title: Virtual Reality Gaming for Exercise and Mindfulness Among Pediatric Cancer Rehabilitation
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Byron Lai, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 300012601; LAIKPRI02012024 (Other Grant/Funding Number: Kaul Pediatric Research Institute Pilot Grant)
Record Dates: First submitted 2024-02-29; First posted 2024-03-07 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: There will be 2 parallel groups, immediate start group and waitlist control group. Once control participants finish the wait period (8 weeks), they will start the intervention (8 weeks). Participants in the immediate start group will start exercise and mindfulness in the hospital and continue the program for 8 weeks outside of the hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Start (Experimental): Program starts in the hospital and lasts for 8 weeks after hospital discharge.
  Interventions: Behavioral: Immediate Start - Virtual Reality
- Waitlist Control (Active Comparator): After 8 weeks after hospital discharge, these participants start the 8 week intervention.
  Interventions: Behavioral: Delayed Start - Virtual Reality

INTERVENTIONS:
Behavioral: Immediate Start - Virtual Reality — Participants will use a Meta Quest virtual reality headset and play video games for exercise and mindfulness. They will start using the headsets in the hospital and then will continue to do so for 8 weeks after hospital discharge.
  Arms: Immediate Start
Behavioral: Delayed Start - Virtual Reality — Participants will receive usual care in the hospital and outside of the hospital for 8 weeks. After the 8 week post-discharge period, participants will use a Meta Quest virtual reality headset and play video games for exercise and mindfulness for an 8 week period.
  Arms: Waitlist Control

SUMMARY:
This study will explore the potential benefits of a virtual reality gaming program that focuses on mindfulness and exercise among pediatric cancer rehabilitation patients. The program will last 8 weeks outside of the hospital. Participants will start immediately in the hospital (immediate start group) or wait 8 weeks after hospital discharge to start the program (waitlist control group).

ELIGIBILITY:
Inclusion Criteria:

* >7 years of age
* medical diagnosis of malignancy or non-malignant condition requiring hematopoietic stem cell transplant or a hospital stay that is anticipated to last for at least 2 weeks
* a caregiver who can assist the child with the study procedures

Exclusion Criteria:

* complete blindness or deafness
* inability to operate the hand-held controllers
* susceptible to motion sickness in virtual reality
* inability to communicate in English

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Physical activity | Daily, starting after consent in the hospital (week 0) and ending after the intervention (intervention week 9)
  Steps per day measured by a tri-axial accelerometer (Fitbit Flex).

SECONDARY OUTCOMES:
Minutes of gameplay | Hospital discharge (approximately week 4), Intervention week 4, and Intervention Week 8.
  Minutes of gameplay measured by the Meta Quest headset.
Global Health | Week 0, ~Week 2 (Post-Transplant), ~Week 4 (hospital discharge), Intervention or Wait Period Week 4, Intervention or Wait Period Week 8.
  National Institutes of Health (NIH) PROMIS Global Health Short Form 7+2 survey. The scale consists of 7 items that are summarized into a single score of overall health. Participants respond to items without a recall period on how they would rate their overall health, quality of life, and their physical, mental, and social health, using a 5-point Likert scale with varying response categories.
Forced Expiratory Volume in the first second (FEV1) | Week 0, ~Week 2 (Post-Transplant), ~Week 4 (hospital discharge), Intervention or Wait Period Week 4, Intervention or Wait Period Week 8.
  FEV1 (Liters) by a Spirometer

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lai B, Chaviano K, Richman JS, Ahmad M, Wright A, Young R, Davis D, Rimmer JH, Madan-Swain A, Chewning JH. Extended Reality Gaming for Exercise and Mindfulness Throughout Pediatric Cancer Rehabilitation: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Dec 23;13:e64879. doi: 10.2196/64879. PMID 39714090